CLINICAL TRIAL: NCT02097225
Title: Phase I Study of AT13387 in Combination With Dabrafenib and Trametinib in Patients With BRAF-Mutant Melanoma and Other Solid Tumors
Brief Title: Onalespib, Dabrafenib, and Trametinib in Treating Patients With BRAF-Mutant Melanoma or Solid Tumors That Are Metastatic or Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug supply issues
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00615; NCI-2014-00615 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CTEP#9557; 14-186; 9557 (Other: Massachusetts General Hospital Cancer Center); 9557 (Other: CTEP); P30CA006516 (NIH); U01CA062490 (NIH); UM1CA186709 (NIH)
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: BRAF V600E Mutation Present; BRAF V600K Mutation Present; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Stage III Cutaneous Melanoma AJCC v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7; Unresectable Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma | interventions — dabrafenib; (2,4-dihydroxy-5-isopropylphenyl)-(5-(4-methylpiperazin-1-ylmethyl)-1,3-dihydroisoindol-2-yl)methanone; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose level -1 (dabrafenib, trametinib, onalespib) (Experimental): Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28, and onalespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  There are four dose levels, plus a fallback dose. Dose escalation begins at dose level 1 (starting dose). Fallback dose level -1 is initiated if more than 1 of 6 subjects in dose level 1 (starting dose) develop DLTs.
  Dose Level -1 (fallback dose):
  * Dabrafenib = 75 mg
  * Trametinib = 1 mg
  * Onalespib = 180 mg/m^2
  Interventions: Drug: Dabrafenib; Other: Laboratory Biomarker Analysis; Drug: Onalespib; Other: Pharmacological Study; Drug: Trametinib
- Dose level 1 (dabrafenib, trametinib, onalespib) (Experimental): Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28, and onalespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  There are four dose levels, plus a fallback dose. Dose escalation begins at dose level 1 (starting dose).
  Dose Level 1 (starting dose):
  * Dabrafenib = 150 mg
  * Trametinib = 1 mg
  * Onalespib = 180 mg/m^2
  Interventions: Drug: Dabrafenib; Other: Laboratory Biomarker Analysis; Drug: Onalespib; Other: Pharmacological Study; Drug: Trametinib
- Dose level 2 (dabrafenib, trametinib, onalespib) (Experimental): Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28, and onalespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  There are four dose levels, plus a fallback dose. Dose escalation begins at dose level 1 (starting dose).
  Dose Level 2:
  * Dabrafenib = 150 mg
  * Trametinib = 2 mg
  * Onalespib = 180 mg/m^2
  Interventions: Drug: Dabrafenib; Other: Laboratory Biomarker Analysis; Drug: Onalespib; Other: Pharmacological Study; Drug: Trametinib
- Dose level 3 (dabrafenib, trametinib, onalespib) (Experimental): Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28, and onalespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  There are four dose levels, plus a fallback dose. Dose escalation begins at dose level 1 (starting dose).
  Dose Level 3:
  * Dabrafenib = 150 mg
  * Trametinib = 2 mg
  * Onalespib = 220 mg/m^2
  Interventions: Drug: Dabrafenib; Other: Laboratory Biomarker Analysis; Drug: Onalespib; Other: Pharmacological Study; Drug: Trametinib
- Dose level 4 (dabrafenib, trametinib, onalespib) (Experimental): Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28, and onalespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  There are four dose levels, plus a fallback dose. Dose escalation begins at dose level 1 (starting dose).
  Dose Level 4:
  * Dabrafenib = 150 mg
  * Trametinib = 2 mg
  * Onalespib = 260 mg/m^2
  Interventions: Drug: Dabrafenib; Other: Laboratory Biomarker Analysis; Drug: Onalespib; Other: Pharmacological Study; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Given PO
  Other Names: BRAF Inhibitor GSK2118436; GSK-2118436; GSK-2118436A; GSK2118436
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Onalespib — Given IV
  Other Names: AT 13387; AT-13387; AT13387
Other: Pharmacological Study — Correlative studies
Drug: Trametinib — Given PO
  Other Names: GSK 1120212; GSK-1120212; GSK1120212; JTP-74057; MEK Inhibitor GSK1120212

SUMMARY:
This phase I trial studies the side effects and best dose of onalespib when given together with dabrafenib and trametinib in treating patients with BRAF-mutant melanoma or solid tumors that have spread to another place in the body (metastatic) or cannot be removed by surgery. Onalespib, dabrafenib, and trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD), toxicity, and safety profile of onalespib (AT13387) given weekly in combination with dabrafenib and trametinib in patients with BRAF-mutant metastatic or unresectable solid tumors.

SECONDARY OBJECTIVES:

I. To obtain preliminary estimates of the objective response rate (ORR) and progression-free survival (PFS) and document the 6-month PFS and 1-year overall survival (OS) of patients with BRAF-mutant metastatic or unresectable melanoma treated with AT13387 given weekly in combination with dabrafenib and trametinib.

II. To describe the pharmacokinetics of treatment with dabrafenib, trametinib, and AT13387.

OUTLINE: This is a dose-escalation study of onalespib. Four dose levels, plus a fallback dose, are specified in the protocol and are summarized below. The trial is based on a standard 3+3 design with dose escalation beginning in dose level 1 (DL1). In a 3+3 design," three patients are initially enrolled into a given dose cohort. If there is no dose limiting toxicity (DLT) observed in any of these subjects, the trial proceeds to enroll additional subjects into the next higher dose cohort. If one subject develops a DLT at a specific dose, an additional three subjects are enrolled into that same dose cohort. Development of DLTs in more than 1 of 6 subjects in a specific dose cohort suggests that the maximum total dose (MTD) has been exceeded, and further dose escalation is not pursued. Fallback dose level -1 is initiated if more than 1 of 6 subjects in dose level 1 (starting dose) develop DLTs.

Patients receive dabrafenib orally (PO) twice daily (BID), trametinib PO once daily (QD) on days 1-28, and onalespib intravenously (IV) over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Dose Level -1 (fallback dose):

* Dabrafenib = 75 mg
* Trametinib = 1 mg
* Onalespib = 180 mg/m^2

Dose Level 1 (starting dose):

* Dabrafenib = 150 mg
* Trametinib = 1 mg
* Onalespib = 180 mg/m^2

Dose Level 2:

* Dabrafenib = 150 mg
* Trametinib = 2 mg
* Onalespib = 180 mg/m^2

Dose Level 3:

* Dabrafenib = 150 mg
* Trametinib = 2 mg
* Onalespib = 220 mg/m^2

Dose Level 4:

* Dabrafenib = 150 mg
* Trametinib = 2 mg
* Onalespib = 260 mg/m^2

After completion of study treatment, patients are followed up at 28 days and every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed, BRAF-mutant (V600E/K) solid tumor (molecularly confirmed using Cobas assay or a comparable Food and Drug Administration [FDA]-approved assay) that is metastatic or unresectable, have received and tolerated prior BRAF or BRAF and MEK inhibitor (BRAF targeted) therapy at full dose or not previously received BRAF targeted therapy, and for which standard curative measures do not exist or are no longer effective

  * If test at Clinical Laboratory Improvement Act (CLIA)-certified laboratory (lab) used a non-FDA approved method, information about the assay must be provided; (FDA approved tests for BRAF V600 mutations in melanoma include: THxID BRAF Detection Kit and Cobas 4800 BRAF V600 Mutation Test)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Prior therapy is allowed; patients may have received any number of prior lines of therapy, including treatment with a BRAF and/or MEK inhibitor
* All prior anti-cancer treatment-related toxicities must be less than or equal to grade 1 according to the Common Terminology Criteria for Adverse Events version 5 (CTCAE version 5.0; National Cancer Institute [NCI], 2017) at the time of enrollment; a notable exception are endocrinopathies caused by immune checkpoint inhibitors that are appropriately treated with medical management (e.g. hormone replacement therapy, anti-diabetic agents)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,200/mcL
* Hemoglobin >= 9 g/dl (patients may be transfused to this level)
* Platelets >= 100,000/mcL
* Total bilirubin < 1.5 x institutional upper limit of normal OR > 1.5 x institutional upper limit of normal allowed if direct bilirubin is within normal range
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Prothrombin time (PT) < 1.3 x upper limit of normal (ULN)
* International normalized ratio (INR) < 1.3 x ULN
* Partial thromboplastin time (PTT) < 1.3 x ULN
* Serum creatinine =< 1.5 mg/dL OR creatinine clearance >= 50 mL/min/1.73 m^2
* Potassium > 3 and < 5.5 mEq/L
* Magnesium > 1.2 and < 2.5 mEq
* Left ventricular >= institutional lower limit of normal (LLN) by echocardiogram (ECHO) ejection fraction
* Women of child-bearing potential must have a negative serum pregnancy test within 14 days prior to randomization and agree to use effective contraception (barrier method of birth control, or abstinence; hormonal contraception is not allowed) from 14 days prior to randomization, throughout the treatment period, and for 4 months after the last dose of study treatment; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately
* Therapeutic level dosing of warfarin can be used with close monitoring of PT/INR by the site; exposure may be decreased due to enzyme induction when on treatment, thus warfarin dosing may need to be adjusted based upon PT/INR; consequently, when discontinuing dabrafenib, warfarin exposure may be increased and thus close monitoring via PT/INR and warfarin dose adjustments must be made as clinically appropriate; prophylactic low dose warfarin may be given to maintain central catheter patency
* Ability to understand and the willingness to sign a written informed consent document
* Able to swallow and retain oral medication, and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels

Exclusion Criteria:

* Patients who received prior systemic anti-cancer therapy (chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy, or vaccine therapy) within the last 3 weeks prior to day 1 of cycle 1; patients are permitted to be on dabrafenib and trametinib standard of care at start of therapy without wash-out period prior to day 1 of cycle 1; dosing will change to protocol determined dose levels on day 1 of cycle 1
* Patients must not have received prior HSP90 inhibitor therapy
* Patients who are receiving any other investigational agents; patients who have taken an investigational drug within 28 days or 5 half-lives (minimum 14 days), whichever is shorter, prior to randomization
* Patients with history of activating RAS mutation positive tumors regardless of interval from current study; however, patients may have concurrent BRAFV600 and RAS mutations in the tumor to be treated with protocol therapy
* Patients must have no clinical evidence of leptomeningeal or brain metastasis causing spinal cord compression that are symptomatic or untreated or not stable for >= 4 weeks (must be documented by imaging) or requiring corticosteroids; subjects on a stable dose of corticosteroids > 1 month or who have been off of corticosteroids for at least 2 weeks can be enrolled with approval of the Cancer Therapy Evaluation Program (CTEP) medical monitor; subjects must also be off of enzyme-inducing anticonvulsants for > 4 weeks
* History of known immediate or delayed hypersensitivity reactions attributed to compounds of similar chemical or biologic composition to AT13387, dabrafenib, or trametinib, or excipients or to dimethyl sulfoxide (DMSO)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active serious infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled diabetes, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued prior to the mother being treated with the study drugs
* Patients known to be human immunodeficiency virus (HIV)-positive patients and on combination antiretroviral therapy are ineligible
* History of another malignancy other than the study indication under this trial within 5 years of study enrollment; does not apply to subjects who underwent successful definitive resection of basal or squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, in situ breast cancer, or other in situ cancers

  * Exception: patients with history of RAS mutation-positive tumors are not eligible regardless of interval from the current study; prospective RAS testing is not required; however, if the results of previous RAS testing are known, they must be used in assessing eligibility
* History of interstitial lung disease or pneumonitis
* History or current evidence/risk of retinal vein occlusion (RVO) or retinal pigment epithelial detachment (RPED):

  * History of RVO or RPED, or predisposing factors to RVO or RPED (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension, diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes)
  * Visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for RVO or RPED such as evidence of new optic disc cupping, evidence of new visual field defects, and intraocular pressure > 21 mm mercury (Hg)
* History or evidence of cardiovascular risk including any of the following:

  * An average of the three most recent QT intervals corrected for heart rate using the Bazett's formula QTcB >= 460 msec
  * History or evidence of current clinically significant uncontrolled arrhythmias (exception: patients with controlled atrial fibrillation for > 30 days prior to randomization are eligible)
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization
  * History or evidence of current >= class II congestive heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
  * Abnormal cardiac valve morphology (>= grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study); subjects with moderate valvular thickening should not be entered on study
  * Prior placement of an implantable defibrillator
  * History of or identification on screening imaging of intracardiac metastases
* No known active infection with hepatitis B virus (HBV), or hepatitis C virus (HCV); patients with chronic or cleared HBV infection and HCV infection are eligible
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited:

  * Other anti-cancer therapy while on study treatment; (note: megestrol [Megace] if used as an appetite stimulant is allowed)
  * Concurrent treatment with bisphosphonates is permitted; however, treatment must be initiated prior to the first dose of study therapy; prophylactic use of bisphosphonates in patients without bone disease is not permitted, except for the treatment of osteoporosis
  * The concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, St. John's wort, kava, ephedra [ma huang], ginkgo biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)
  * Current use of a prohibited medication; patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A or CYP2C8 are ineligible; current use of, or intended ongoing treatment with: herbal remedies (e.g., St. John's wort), or strong inhibitors or inducers of P-glycoprotein (Pgp) or breast cancer resistance protein 1 (Bcrp1) should also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-05-29 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Sullivan, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Mooradian MJ, Cleary JM, Giobbie-Hurder A, Darville LNF, Parikh A, Buchbinder EI, Cohen JV, Lawrence DP, Shapiro GI, Keer H, Chen HX, Ivy SP, Smalley KSM, Koomen JM, Sullivan RJ. Dose-escalation trial of combination dabrafenib, trametinib, and AT13387 in patients with BRAF-mutant solid tumors. Cancer. 2023 Jun 15;129(12):1904-1918. doi: 10.1002/cncr.34730. Epub 2023 Apr 11. PMID 37042037

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level -1: Dabrafenib = 75 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2: Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28, and onalespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  There are four dose levels, plus a fallback dose. Dose escalation begins at dose level 1 (starting dose). Fallback dose level -1 is initiated if more than 1 of 6 subjects in dose level 1 (starting dose) develop DLTs.
  * Dose Level -1 (fallback dose):
  * Dabrafenib = 75 mg
  * Trametinib = 1 mg
  * Onalespib = 180 mg/m2
  Dabrafenib: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Onalespib: Given IV
  Pharmacological Study: Correlative studies
  Trametinib: Given PO
- Dose Level 1: Dabrafenib = 150 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2: Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28, and onalespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  There are four dose levels, plus a fallback dose. Dose escalation begins at dose level 1 (starting dose).
  * Dose Level 1 (starting dose):
  * Dabrafenib = 150 mg
  * Trametinib = 1 mg
  * Onalespib = 180 mg/m2
  Dabrafenib: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Onalespib: Given IV
  Pharmacological Study: Correlative studies
  Trametinib: Given PO
- Dose Level 2: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 180 mg/m2: Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28, and onalespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  There are four dose levels, plus a fallback dose. Dose escalation begins at dose level 1 (starting dose).
  * Dose Level 2:
  * Dabrafenib = 150 mg
  * Trametinib = 2 mg
  * Onalespib = 180 mg/m2
  Dabrafenib: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Onalespib: Given IV
  Pharmacological Study: Correlative studies
  Trametinib: Given PO
- Dose Level 3: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 220 mg/m2: Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28, and onalespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  There are four dose levels, plus a fallback dose. Dose escalation begins at dose level 1 (starting dose).
  * Dose Level 3:
  * Dabrafenib = 150 mg
  * Trametinib = 2 mg
  * Onalespib = 220 mg/m2
  Dabrafenib: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Onalespib: Given IV
  Pharmacological Study: Correlative studies
  Trametinib: Given PO
- Dose Level 4: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 260 mg/m2: Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28, and onalespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  There are four dose levels, plus a fallback dose. Dose escalation begins at dose level 1 (starting dose).
  * Dose Level 4:
  * Dabrafenib = 150 mg
  * Trametinib = 2 mg
  * Onalespib = 260 mg/m2
  Dabrafenib: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Onalespib: Given IV
  Pharmacological Study: Correlative studies
  Trametinib: Given PO
Period: Dose Level 1
Arm/Group | Dose Level -1: Dabrafenib = 75 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 1: Dabrafenib = 150 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 2: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 180 mg/m2 | Dose Level 3: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 220 mg/m2 | Dose Level 4: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 260 mg/m2
Started | 0 | 3 | 0 | 0 | 0
Completed | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Level 2
Arm/Group | Dose Level -1: Dabrafenib = 75 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 1: Dabrafenib = 150 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 2: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 180 mg/m2 | Dose Level 3: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 220 mg/m2 | Dose Level 4: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 260 mg/m2
Started | 0 | 0 | 4 | 0 | 0
Completed | 0 | 0 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Level 3
Arm/Group | Dose Level -1: Dabrafenib = 75 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 1: Dabrafenib = 150 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 2: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 180 mg/m2 | Dose Level 3: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 220 mg/m2 | Dose Level 4: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 260 mg/m2
Started | 0 | 0 | 0 | 6 | 0
Completed | 0 | 0 | 0 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Level 4
Arm/Group | Dose Level -1: Dabrafenib = 75 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 1: Dabrafenib = 150 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 2: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 180 mg/m2 | Dose Level 3: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 220 mg/m2 | Dose Level 4: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 260 mg/m2
Started | 0 | 0 | 0 | 0 | 9
Completed | 0 | 0 | 0 | 0 | 8
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: No participants were enrolled into fallback Dose Level -1 because Dose Level -1 is only initiated if more than 1 of 6 subjects in dose level 1 (starting dose) develop DLTs.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level -1: Dabrafenib = 75 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 1: Dabrafenib = 150 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 2: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 180 mg/m2 | Dose Level 3: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 220 mg/m2 | Dose Level 4: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 260 mg/m2 | Total
Number analyzed (Participants) | 0 | 3 | 4 | 6 | 9 | 22
Age, Continuous [Median (Full Range); unit: years] |  | 51.0 [51.0 to 66.0] | 66.5 [58.0 to 69.0] | 54.0 [43.0 to 68.0] | 58.0 [37.0 to 75.0] | 57.5 [37.0 to 75.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 4 | 5 | 13
  Male | 0 | 2 | 1 | 2 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 3 | 4 | 6 | 8 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is a simple measure of functional status. Scores range from 0 to 5, where higher scores indicate lower functional status. Eligibility criteria for this trial allowed for scores 0 or 1.
  Score 0 = Fully active, able to carry on all pre-disease performance without restriction.
  Score 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    Score 0 | 0 | 0 | 0 | 3 | 4 | 7
    Score 1 | 0 | 3 | 4 | 3 | 5 | 15
Months since diagnosis at time of study enrollment [Median (Full Range); unit: months] |  | 7.8 [6.0 to 10.5] | 19.2 [9.1 to 32.5] | 68.8 [14.5 to 346.0] | 18.9 [6.1 to 57.8] | 19.7 [6.0 to 346.0]
Disease Histology [Count of Participants; unit: Participants]
  Adenocarcinoma of colon |  | 2 | 4 | 2 | 4 | 12
  Metastatic melanoma |  | 1 | 0 | 2 | 3 | 6
  Adenocarcinoma of lung |  | 0 | 0 | 0 | 1 | 1
  Epithelioid sarcoma |  | 0 | 0 | 1 | 0 | 1
  Anaplastic thyroid carcinoma |  | 0 | 0 | 0 | 1 | 1
  Adenocarcinoma, Not otherwise specified |  | 0 | 0 | 1 | 0 | 1
Prior Therapy Received [Count of Participants; unit: Participants] — Participants may have had more than one therapy type.
  Participants
    Chemotherapy, not otherwise specified |  | 0 | 0 | 1 | 1 | 2
    Chemotherapy, multiple agents systemic |  | 3 | 4 | 4 | 8 | 19
    Chemotherapy, single agent systemic |  | 1 | 1 | 2 | 3 | 7
    Chemotherapy, non-cytotoxic |  | 0 | 0 | 1 | 0 | 1
    Immunotherapy |  | 1 | 1 | 3 | 3 | 8
    Limited Radiation Therapy |  | 1 | 0 | 1 | 3 | 5
    Radiation Therapy, not otherwise specified |  | 1 | 0 | 1 | 1 | 3
    Surgery |  | 3 | 4 | 6 | 9 | 22
    Vaccine therapy |  | 0 | 0 | 1 | 0 | 1
    Prior therapy, not otherwise specified |  | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Dabrafenib
Description: Maximum tolerated dose is defined as the highest dose level at which 0 or 1 of six patients has experienced a dose limiting toxicity (DLT) within 28 days after start of treatment. Toxicities will be graded according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0. Participant enrollment occurred from July 2015 to June 2018, spanning Dose Levels 1-4.
  * Dose Level 1 (starting dose):
    * Dabrafenib = 150 mg
    * Trametinib = 1 mg
    * Onalespib = 180 mg/m2
  * Dose Level 2:
    * Dabrafenib = 150 mg
    * Trametinib = 2 mg
    * Onalespib = 180 mg/m2
  * Dose Level 3:
    * Dabrafenib = 150 mg
    * Trametinib = 2 mg
    * Onalespib = 220 mg/m2
  * Dose Level 4:
    * Dabrafenib = 150 mg
    * Trametinib = 2 mg
    * Onalespib = 260 mg/m2
Time Frame: 28 days after start of treatment
Measure: Number; unit: mg
Groups:
- Treatment (Dabrafenib, Trametinib, Onalespib): Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28, and onalespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Four dose levels, plus a fallback dose, are summarized in the table below. Dose escalation begins at dose level 1 (starting dose).
  * Dose Level -1:
    * Dabrafenib = 75 mg
    * Trametinib = 1 mg
    * Onalespib = 180 mg/m2
  * Dose Level 1 (starting dose):
    * Dabrafenib = 150 mg
    * Trametinib = 1 mg
    * Onalespib = 180 mg/m2
  * Dose Level 2:
    * Dabrafenib = 75 mg
    * Trametinib = 1 mg
    * Onalespib = 180 mg/m2
  * Dose Level 3:
    * Dabrafenib = 150 mg
    * Trametinib = 2 mg
    * Onalespib = 220 mg/m2
  * Dose Level 4:
    * Dabrafenib = 150 mg
    * Trametinib = 2 mg
    * Onalespib = 260 mg/m2
  Dabrafenib: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Onalespib: Given IV
  Pharmacological Study: Correlative studies
  Trametinib: Given PO
Arm/Group | Treatment (Dabrafenib, Trametinib, Onalespib)
Number analyzed (Participants) | 21
mg | 150

2. Primary Outcome: Maximum Tolerated Dose of Trametinib
Description: as for outcome 1
Time Frame: 28 days after start of treatment
Measure: Number; unit: mg
Arm/Group | Treatment (Dabrafenib, Trametinib, Onalespib)
Number analyzed (Participants) | 18
mg | 2

3. Primary Outcome: Maximum Tolerated Dose of Onalespib
Description: as for outcome 1
Time Frame: 28 days after start of treatment
Measure: Number; unit: mg/m2
Arm/Group | Treatment (Dabrafenib, Trametinib, Onalespib)
Number analyzed (Participants) | 8
mg/m2 | 260

4. Primary Outcome: Number of Dose Limiting Toxicities While Determining Maximum Tolerated Dose
Description: Dose limiting toxicities (DLTs) are at least possibly related to study treatment and graded according to the Common Toxicity Criteria for Adverse Events (CTCAE) v5.0:
  * any grade 4 toxicity
  * grade 3 (or grade 2 intolerable) non-hematologic toxicity (including fatigue lasting >1 week or that requires hospitalization)
  * grade 3 or higher hematologic toxicity with complications (e.g., thrombocytopenia with bleeding, neutropenia with fever)
  * toxicity that lead to missing a dose of onalespib or >25% of dabrafenib/trametinib in the first cycle
  The following grade 3 toxicities are not considered DLTs:
  * cutaneous squamous cell carcinoma or keratoacanthoma
  * nausea, vomiting, or diarrhea persisting </= 72 hours with maximum supportive care
  * electrolyte events that resolve with replacement within 24 hours
  * any grade lymphopenia
  * lab abnormalities that return to baseline within 7 days: elevated bilirubin, AST, ALT, cholesterol, amylase, lipase, creatinine, hypertriglyceridemia
Time Frame: 28 days after start of treatment (1 cycle)
Measure: Number; unit: dose limiting toxicities
Groups:
- Dose Level 1: Dabrafenib = 150 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2: Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28, and onalespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Four dose levels, plus a fallback dose, are summarized in the table below. Dose escalation begins at dose level 1 (starting dose).
  *Dose Level 1 (starting dose):
  * Dabrafenib = 150 mg
  * Trametinib = 1 mg
  * Onalespib = 180 mg/m2
  Dabrafenib: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Onalespib: Given IV
  Pharmacological Study: Correlative studies
  Trametinib: Given PO
Arm/Group | Dose Level 1: Dabrafenib = 150 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 2: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 180 mg/m2 | Dose Level 3: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 220 mg/m2 | Dose Level 4: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 260 mg/m2
Number analyzed (Participants) | 3 | 4 | 6 | 8
dose limiting toxicities
  Grade 3 toxicity | 0 | 0 | 5 | 1
  Grade 4 toxicity | 0 | 0 | 0 | 0

5. Secondary Outcome: Objective Response Rate
Description: Objective response rate is defined as the number of participants with complete response or partial response as their best response to therapy assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
  * Complete response (CR) = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial response (PR) = At least a 30% decrease in the sum of longest diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Dabrafenib = 150 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 2: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 180 mg/m2 | Dose Level 3: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 220 mg/m2 | Dose Level 4: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 260 mg/m2
Number analyzed (Participants) | 3 | 4 | 6 | 8
Participants
  Complete response (CR) | 0 | 0 | 0 | 0
  Partial response (PR) | 0 | 0 | 2 | 0

6. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progressive disease assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1, or death, whichever occurs first.
  Progressive disease (PD) = At least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the baseline sum of diameters. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progressions.
Time Frame: up to 9 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Dose Level 1: Dabrafenib = 150 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 2: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 180 mg/m2 | Dose Level 3: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 220 mg/m2 | Dose Level 4: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 260 mg/m2
Number analyzed (Participants) | 3 | 4 | 6 | 8
months | 1.6 [0.9 to 1.7] | 1.5 [0.6 to 3.6] | 3.9 [1.8 to 9.2] | 2.7 [1.5 to 3.8]

7. Secondary Outcome: Progression-free Survival at 6 Months
Description: Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progressive disease assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1, or death, whichever occurs first. PFS at 6 months will report the number of participants without progression at 6 months after starting treatment.
  Progressive disease (PD) = At least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the baseline sum of diameters. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progressions.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Dabrafenib = 150 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 2: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 180 mg/m2 | Dose Level 3: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 220 mg/m2 | Dose Level 4: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 260 mg/m2
Number analyzed (Participants) | 3 | 4 | 6 | 8
Participants | 0 | 0 | 2 | 2

8. Secondary Outcome: Overall Survival at 1 Year
Description: Overall survival (OS) is defined as the time from start of treatment to death from any cause. OS at 1 year will report the number of participants alive at 1 year after starting treatment.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Dabrafenib = 150 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 2: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 180 mg/m2 | Dose Level 3: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 220 mg/m2 | Dose Level 4: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 260 mg/m2
Number analyzed (Participants) | 3 | 4 | 6 | 8
Participants | 0 | 0 | 1 | 3

9. Other Pre Specified Outcome: Pharmacokinetics of Dabrafenib, Trametinib, and Onalespib Combination
Description: Pharmacokinetics (PKs) represents the absorption, distribution, metabolism, and elimination of study drugs from the body.
  PKs for this study are reported a Area Under the Curve (AUC), which is estimated using the trapezoidal rule based on the average drug concentrations in blood samples, specifically blood plasma, at 1 hour immediately after study drug infusion.
  AUC gives insight into the extent of exposure to a drug and its clearance rate from the body.
Time Frame: 1 hour immediately after Cycle 1, Day 1 infusion
Population: There were 18 out of 21 total evaluable patients had blood samples analyzed on Cycle 1 Day 1.
Measure: Median (Full Range); unit: ng*hr/mL
Arm/Group | Dose Level 1: Dabrafenib = 150 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 2: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 180 mg/m2 | Dose Level 3: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 220 mg/m2 | Dose Level 4: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 260 mg/m2
Number analyzed (Participants) | 3 | 3 | 6 | 6
ng*hr/mL | 357 [182 to 374] | 344 [210 to 348] | 395 [312 to 502] | 448 [362 to 2310]

ADVERSE EVENTS:
Time Frame: Up to approximately 4.5 years, starting from the day 1 of dosing throughout post-treatment follow-up.
Arm/Group | Dose Level 1: Dabrafenib = 150 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 | Dose Level 2: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 180 mg/m2 | Dose Level 3: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 220 mg/m2 | Dose Level 4: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 260 mg/m2
All-Cause Mortality (participants affected / at risk) | 3/3 | 4/4 | 6/6 | 7/8
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 0/6 | 2/8
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 6/6 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: Dabrafenib = 150 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 (N=3) | Dose Level 2: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 180 mg/m2 (N=4) | Dose Level 3: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 220 mg/m2 (N=6) | Dose Level 4: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 260 mg/m2 (N=8)
Investigations - Other, specify (Investigations) | 1 | 1 | 0 | 2 — death due to disease progression
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Infections and infestations Other, specify (Infections and infestations) | 0 | 0 | 0 | 1 — line infection
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: Dabrafenib = 150 mg, Trametinib = 1 mg, Onalespib = 180 mg/m2 (N=3) | Dose Level 2: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 180 mg/m2 (N=4) | Dose Level 3: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 220 mg/m2 (N=6) | Dose Level 4: Dabrafenib = 150 mg, Trametinib = 2 mg, Onalespib = 260 mg/m2 (N=8)
Thromboembolic Event (Vascular disorders) | 1 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 1
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Gait Disturbance (General disorders) | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Pneumonia
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Pain, unspecified (General disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Alkaline Phosphatase Increased (Investigations) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
White Blood Cell Decreased (Investigations) | 0 | 0 | 2 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 1
Colonic Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT02097225/Prot_SAP_000.pdf